



**CONSENT FORM** 

| Study Number: | 2019003AN | IRAS Number: 261698 |
|---------------|-----------|---------------------|

Individual Participant Identification Number for this trial:

Title of Study: Can continuous non-invasive monitoring improve stability of intraoperative blood pressure

(iSTABILISE)

Name of Researcher: Dr William Rook

| | | Particip | pant to initial box |
|---|---|---|---|
| 1. | I confirm that I have read the information sheet date<br>above study. I have had the opportunity to consider<br>had these answered satisfactorily. | , | |
| 2. | I understand that my participation is voluntary and t<br>without giving any reason, without my medical care | • | |
| 3. | I understand that relevant sections of my medical not<br>the study may be looked at by individuals from regular<br>from the NHS Trust, where it is relevant to my taking<br>these individuals to have access to my records. | ulatory authorities or | |
| 4. | I understand that the information collected about me<br>other related research in the future and may be sha | • • | |
| 5. | I agree to take part in the above study. | | |
| 6. | 6. If you wish to be informed of the study results please write your contact details here: | | |
| | e of Participant Date felement | Signature | |

iStabilise Consent Form - IRAS ID: 261698

Date

V1.1 06-06-19

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.

Signature

taking consent



iStabilise Consent Form – IRAS ID: 261698

V1.1 06-06-19

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.